CLINICAL TRIAL: NCT00852982
Title: Exercise - Effects on Health Related Quality of Life, Cardiovascular Risk Factors, and Cellular Functions With Respect to Glucose Metabolism, in Type 2 Diabetes Mellitus, Impaired Glucose Tolerance and in Healthy Individuals.
Brief Title: Exercise Effects on Cardiovascular Risk Factors, Quality of Life, Muscle Function in Type 2 Diabetes and Healthy Persons
Acronym: SMIDIG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Juleen Zierath , Professor, Dep. of molecular medicine and surgery, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALF 2006 03 25
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2009-03-02 (Estimated); Status verified 2009-02

CONDITIONS: Type 2 Diabetes; Impaired Glucose Tolerance
Keywords: Exercise; Risk factors; Primary health care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Five hours of Nordic walking per week, during four months
  Interventions: Behavioral: Exercise
- Control (No Intervention): Control group asked not to alter lifestyle during study
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Nordic walking, with walking poles, five hours per week during four months

SUMMARY:
A sedentary lifestyle is known to be a risk factor to developing type 2 diabetes. The aim of this study was to determine the effects of adding regular Nordic walking to daily physical activity. Effects on quality of life, cardiovascular risk factors and functions in muscle cells will be determined.

DETAILED DESCRIPTION:
Regular physical activity is known to have a beneficial effect on several factors affecting the risk of developing cardiovascular disease and type 2 diabetes. Implementing and maintaining changes of lifestyle is, however, known to be difficult. In this study we wished to investigate the effects of an exercise intervention that is feasible to most people with type 2 diabetes or at risk of developing that disease. The intervention was Nordic walking (with walking poles) for five hour per week, during four months. We chose to determine effects on health related quality of life, clinical parameters related to body weight/body composition, blood pressure, glucose metabolism, insulin resistance, blood lipids, oxygen uptake and physiological effects in skeletal muscle cells related to glucose metabolism.

On inclusion and after four months the participants were therefore subject to clinical measurements, blood samples, maximal oxygen uptake tests on an ergometer cycle and muscle biopsies at inclusion and after four months of participation. They also answered an extensive questionnaire focusing on health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* BMI>25

Exclusion Criteria:

* Physical impairment
* Symptomatic angina pectoris
* Insulin treatment

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
HbA1c | at inclusion and after four months

SECONDARY OUTCOMES:
waist circumference | at inclusion and after four months

CONTACTS AND LOCATIONS:
Overall Officials: Juleen Zierath, Professor, Principal Investigator — Dep. of molecular medicine and surgery, Karolinska Institutet
Locations (1):
- Primary health care center, Stockholm, Sweden

REFERENCES:
- [Derived] Osler ME, Fritz T, Caidahl K, Krook A, Zierath JR, Wallberg-Henriksson H. Changes in gene expression in responders and nonresponders to a low-intensity walking intervention. Diabetes Care. 2015 Jun;38(6):1154-60. doi: 10.2337/dc14-2606. Epub 2015 Mar 20. PMID 25795414
- [Derived] Fritz T, Caidahl K, Osler M, Ostenson CG, Zierath JR, Wandell P. Effects of Nordic walking on health-related quality of life in overweight individuals with type 2 diabetes mellitus, impaired or normal glucose tolerance. Diabet Med. 2011 Nov;28(11):1362-72. doi: 10.1111/j.1464-5491.2011.03348.x. PMID 21658122